CLINICAL TRIAL: NCT03728387
Title: The Validity, Reliability and Responsiveness of the Fullerton Advanced Balance (FAB-T) Scale in Patients With Osteoarthritis
Brief Title: The Validity, Reliability and Responsiveness of the Fullerton Advanced Balance Scale in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sevim Öksüz, Asst. Prof., Eastern Mediterranean University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2018-0203
Record Dates: First submitted 2018-10-26; First posted 2018-11-02 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Osteo Arthritis Knee; Exercise; Balance
Keywords: osteoarthritis; exercise; balance
MeSH Terms: conditions — Motor Activity; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osteoarthritis and clinical pilates exercise (Experimental): 34 volunteer individuals who will be randomly choosen among 84 individuals will be given a 6-week exercise training program. According to this 6 week program, individuals will be admitted to the exercise training program for 45-60 minutes with a physiotherapist for 3 days in a week. The exercise program will consist of a warm-up, a strength training and a cool-down section.
  Interventions: Other: Clinical Pilates Exercise

INTERVENTIONS:
Other: Clinical Pilates Exercise — All evaluations of the individuals included in the study will be done by the physiotherapist.. For the second evaluation the same individuals will be visited by the same physiotherapist at least 7 days after the first evaluation and only the FAB-T scale will be applied. 34 volunteer individuals who will be randomly choosen among 84 individuals will be given a 6-week exercise training program. According to this 6 week program, individuals will be admitted to the exercise training program for 45-60 minutes with a physiotherapist for 3 days in a week. The exercise program will consist of a warm-up, a strength training and a cool-down section. Various exercise methods (clinical pilates exercises) and tools will be utilized to improve balance and mobility. Third assessment of FAB-T will be applied only to individuals participating in the 6-week exercise training program.

SUMMARY:
The primary aim of our study is to evaluate the validity and reliability of the Fullerton Advanced Balance (FAB-T) scale in individuals with osteoarthritis. The secondary aim of this study is to evaluate the responsiveness of the FAB-T scale to change in patients with osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common joint disorder (1). OA is seen 7 times more than rheumatoid artritis. It is the most important cause of disability seen with advanced age (1). It's a degenerative joint disease, usually associated with progressing age and characterized by biochemical and morphological changes in the synovial membrane and joint capsule, erosion of the joint cartilage, hypertrophy of the joint edges, subchondral sclerosis (2).

OA, an important public health problem, affects the knee joint most frequently (3). While the most important risk factor is age, there are many other risk factors such as race, sex, obesity, genetics and trauma. In osteoarthritis; joint is damaged due to the imbalance between formation and destruction. It causes progressive joint damage, pain, physical disability, and psychological disorders (4). The clinical characteristics of OA include pain, stiffness, limitation of motion, crepitation, varying degrees of inflammation and effusion, disability, functional disability, loss of daily living activities, deterioration in quality of life. (4,5). Pain is diminished by increased resting and alleviated by movement but advanced stages may also include resting pain and night pain. (6) In painful, swollen joints; loss of function is inevitable. The loss of function is specific to the site which is being involved. In knee OA, difficulty in squatting and climbing stairs, walking distance reduction and fatigue, antalgic gait can be seen (7). These complaints are often associated with instability. With increasing age, the frequency of OA also increases. The presence of knee OA in addition to the complications associated with aging especially affects the quality of life negatively. In addition to the physiological effects of advancing age; pain, functional restriction, loss of proprioception and instability due to knee OA may lead to a decrease in balance and, consequently, to falls, which may lead to undesirable outcomes. The determination of the balance problems in OA patients is also important in planning the treatment protocol to be given and also in evaluating the effectiveness of the treatment. There are valid and reliable scales in Turkish language which assess balance.

However, validity and reliability specific to the disease are also important for doing the assessment safeley in that population.

The Fullerton Advanced Balance Scale (FAB) was developed by Debbie Rose in 2006 to evaluate patients with a high risk of falling. The test uses dynamic and static equilibrium in different situations to determine balance problems in the elderly. The test has 10 parameters. These are: feet adjacent and eyes closed standing, reaching out forward to reach a shoulder-length object, turning in right and left directions in 360 degrees, stepping and passing over a 15.24 cm-length stair, tandem march, standing on one leg, eyes closed standing on the foam, double feet bounce, walking with head turning, reactive postural control. In this scale, which is scored between 0-40, a score between 0 and 4 is given for each item (8).

According to the power analysis,a total number of 84 knee osteoarthritis patients, aged between 40 and 65 years of age will be included in the study. Individuals will be given written and oral information about the study and their written approvals will be obtained. * The Turkish version of the Fullerton Advanced Balance Scale (FAB) was obtained with permission from Debbie Rose who developed the scale and it is used on the elderly before. Study pattern: Familiarization will be made to the physiotherapists before the study. Information about the all scales will be given in detail with practical application. The study will be performed on 3 different days and by a single physiotherapist. 1st Evaluation: All evaluations of the individuals included in the study will be done by the physiotherapist (sociodemographic evaluations, implementation of FAB-T and other balance scales). In addition, to determine the acceptability of the FAB-T scale, the time during the FAB-T application will be recorded. 2nd Evaluation: The same individuals will be visited by the same physiotherapist at least 7 days after the first evaluation and only the FAB-T scale will be applied. 3rd Evaluation: After 6 weeks of treatment, the FAB-T scale will be applied to all individuals included in the study. The first two evaluations will be made for all participants. After the second evaluation is completed, 34 volunteer individuals who will be randomly choosen among 84 individuals will be given a 6-week exercise training program. According to this 6 week program, individuals will be admitted to the exercise training program for 45-60 minutes with a physiotherapist for 3 days in a week. The exercise program will consist of a warm-up, a strenght training and a cool-down section. Various exercise methods (clinical pilates exercises) and tools will be utilized to improve balance and mobility. Third assessment will be applied only to individuals participating in the 6-week exercise training program. With the study design, the reliability of testing and retesting ability of the FAB-T scale, its validity with respect to its correlation with other balance scales, its acceptability with the application period and its sensitivity to change after 6 weeks of treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with knee osteoarthritis II-III level according to the results of radiological evaluation by Kellgren and Lawrence
* Individuals aged between 40 and 65 years
* Individuals who have pain in his/her either of the knees in 3 month period and who have a VAS score of 3 or more
* Individuals who can walk 10 meters independently (with or without ancillary device)

Exclusion Criteria:

* Individuals with Body Mass Index 35 and above
* Individuals with a history of surgery or injury involving the lower limb within the last 1 year (knee / hip endoprosthesis, post-fracture surgery, menisectomy, etc.)
* Individuals who received hyaluronic acid or corticosteroid injections in the last year
* People with severe eyesight, hearing disabilities Individuals with neurological deficit or disorder
* Individuals with regular exercise habits in the last 6 months
* Individuals with inflammatory rheumatic diseases.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Fullerton Advanced Balance Scale (FAB-T): | Change will be assessed from the baseline at 1 week and 6th week.
  It is a test that determines the functional balance state of individuals. The test has 10 parameters. These are: feet adjacent and eyes closed standing, reaching out forward to reach a shoulder-length object, 360 degrees of turning in right and left directions, stepping and passing over a 15.24 cm-long stair, tandem march, standing on one leg, eyes closed staying on the foam, double feet bounce, walking with head turning, reactive postural control. In this scale, which is scored between 0-40, a score between 0 and 4 is given for each item (8).

SECONDARY OUTCOMES:
Socio-demographic evaluations | it will be recorded at the beginning
  The sociodemographic variables such as age, gender, body mass index (BMI), marital status, education level and occupational status will be recorded. It will also be questioned whether there are problems with the use of auxiliary devices, problems of loss of balance, activities that individual lost balance, whether if they experience falling problems, for how many years they have been experiencing this problem, whether if there is a fall or fall injury.
Berg Balance Test | First evaluation will be applied on the first day and after 6 weeks.
  is a routine test used in daily life, consisting of evaluation of 14 activities, requiring both dynamic and static balance. If the total score is between 0 and 20, there is a high risk of falling, between 21 and 40 there is a moderate risk of falling, between 41-56 there is a low risk of falling(9).
The Timed Up & Go (TUG) Test: | First evaluation will be applied on the first day and after 6 weeks.
  TUG is a frequently used balance test to assess the functional mobility of individuals. It was developed by Podsiadlo and Richardson in 1991. Test measures the speed during many functional maneuvers such as standing up, walking, turning and sitting. In the test, the person is asked to get up from the chair, to walk for 3 meters with his/her own normal speed, to walk back and to sit on the chair and the time is recorded in seconds (sec). A shorter time indicates better balance and mobility. The starting position should be standardized. It is performed 3 times and the average value is recorded (10).
Single Leg Stance Test | First evaluation will be applied on the first day and after 6 weeks.
  1. Single Leg Stance Test on Hard Ground: the patient is asked to flex the knee with eyes open, hands on the hips, feet naked, and the hip in neutral position. The time is started as soon as the foot is removed from the ground and recorded in seconds. The patient is asked to stand on one foot until the arms move or until the foot is dropped on the floor or until the time reaches 60 sec. For each foot, 3 attempts are made and the average time for each foot is recorded. Rest is allowed between attempts.
  2. Single Leg Stance Test on Foam Ground: Eyes open, hands on the hips, feet naked, hip in neutral position on the foam, participant is required to flex a knee. The patient is asked to stand on one foot until the arms move or until the foot is dropped on the floor or until the time reaches 60 sec. For each foot, 3 attempts are made and the average time for each foot is recorded. Rest is allowed between attempts.
Push and Release Test | First evaluation will be applied on the first day and after 6 weeks.
  While the patient is in the standing position with the eyes open, the physiotherapist stands behind the person and places his/her hand on the person's scapula and participant leans backwards to push the hand of the physiotherapist. The physiotherapist flexes the elbows to allow back movement of the body and supports the person's weight with his/her hands. When a person's shoulders and hips are in a fixed position just behind the heels, the physiotherapist suddenly raises participant's hands. Scoring is based on the response of the individual in trying to regain balance. Scoring: 0. = It gains balance independently with 1 step in normal length and width, 1. = Takes two or three small steps backwards, but independently gains equilibrium, 2. = Takes four or more steps backwards, but independently restores balance, 3 . = Takes the step, but need help to prevent he/she from falling, 4. = falls off without taking a step or can't stop without help (13).
30 Seconds Sit and Stand Up Test | First evaluation will be applied on the first day and after 6 weeks.
  For proximal muscle strength of the lower extremity and endurance, this test is valid and reliable for adults. In his/her starting position, the person sits on an armless armchair with his back straight, arms crossed in front of the chest and feet on the ground. With the starting of the measument, the person takes the sitting position from a full standing position and the exact numbers of standing uıp within 30 seconds are recorded. Less than 10 repetitions in 30 seconds show lower extremity muscle weakness. The test is performed once (14).
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index: | First evaluation will be applied on the first day and after 6 weeks.
  consists of 24 questions and is divided into 3 subgroups. WOMAC subgroups consisted of 5 pain-related questions, 2 stiffness-related questions, 17 physical function-related problems. In WOMAC assessment, each question is between 0-4 points. Subgroups are evaluated among themselves. According to this, the subgroup of pain is 0-20 points, the stiffness / rigidity is 0-8 points and the physical function subgroup is 0-68 points. During the evaluation of pain, the severity of pain in the last 24 hours is questioned. For stiffness / rigidity sub-parameters, first; the feeling of stiffness is defined and the joint stiffness felt within the last 24 hours in the evaluated joint is questioned. For physical function score, 17 activities that is being challenging for the participant due to arthralgia in the joint is being questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Ender Angın, PhD, Study Director — Eastern Mediterranen University; Berkiye Kırmızıgil, PhD, Principal Investigator — Eastern Mediterranean University; Gozde Iyigun, PhD, Principal Investigator — Eastern Mediterranean University; Sevim Oksuz, PhD, Principal Investigator — Eastern Mediterranean University; Unal Deger, MSc, Principal Investigator — Eastern Mediterranean University; Filiz Can, Prof, Principal Investigator — Hacettepe University; Levent Eker, MD, Principal Investigator — Eastern Mediterranean University; Debra J. Rose, PhD, Principal Investigator — California State University
Locations (1):
- Eastern Mediterranen University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided